CLINICAL TRIAL: NCT04710225
Title: Does Anesthetic Technique Affect Pneumatic Tourniquet Pressures in Upper Limb Fracture Surgery? A Comparison of General Anesthesia and Axillary Brachial Plexus Block
Brief Title: Does Anesthetic Technique Affect Pneumatic Tourniquet Pressures in Upper Limb Fracture Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Bahattin Tuncali, Associate professor, MD, Baskent University Ankara Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KA19/326
Record Dates: First submitted 2021-01-10; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Initial Systolic Blood Pressure (mmHg); Arterial Occlusion Pressure (mmHg); Tourniquet Time (Minutes); Quality of Bloodless Surgical Field (4 Point Scale); Initial Tourniquet Pressure (mmHg); Maximal Systolic Blood Pressure (mmHg); Maximal Tourniquet Pressure (mmHg)
Keywords: Pneumatic tourniquet; Pressure; Upper extremity; General anesthesia; Axillary brachial plexus block.
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (General anesthesia group) (Active Comparator): Upper limb fracture surgery will be performed with the aid of pneumatic tourniquet. General anesthesia will be induced with intravenous (IV) thiopental sodium and fentanyl.
  Rocuronium will be used as the neuromuscular blocking agent. Endotracheal tube will be placed and anesthesia will be maintained with sevoflurane and IV fentanyl while the lungs were ventilated with O2-N2O (50-50%) to achieve an EtCO2 at 30-35 mm Hg.
  Interventions: Procedure: Upper limb fracture surgery and arterial occlusion pressure (AOP) estimation based tourniquet pressure (TP) setting
- Group 2 (Multiple injection axillary block group) (Active Comparator): Multiple injection axillary block will be performed with the aid of a nerve stimulator. When the slight twitching of the motor response from the relevant muscles is achieved (at 0.4 mA, 2Hz, 0.1 ms) % 18-20 ml of Bupivacaine 0.5 (90-100 mg) will be injected.
  Interventions: Procedure: Upper limb fracture surgery and arterial occlusion pressure (AOP) estimation based tourniquet pressure (TP) setting

INTERVENTIONS:
Procedure: Upper limb fracture surgery and arterial occlusion pressure (AOP) estimation based tourniquet pressure (TP) setting — Upper limb fracture surgery will be performed with the aid of a pneumatic tourniquet.
  The cuff (11 cm) of the tourniquet will be placed around the arm with the distal edge 5 cm above the olecranon. AOP estimation formula according to initial systolic blood pressure (SBP) and Tissue Padding Coefficient (KTP) values (AOP= [SBP+10]/KTP) from a list (Table 1) will be used to calculate AOP (17). After calculation of AOP, a safety margin of 20 mmHg will be added to AOP to determine the TP (TP=AOP+20 mm Hg). Exsanguination of the limb will be provided with an Esmarch bandage and the cuff will be inflated to the predetermined TP. TP will be manually raised in response to each 10 mmHg increase in SBP during the surgical procedure.

SUMMARY:
In pneumatic tourniquet applications, the use of an individualized, lowest-effective tourniquet pressure (TP) has been recommended, in order to avoid pressure related complications. The aim of this study is to compare the effects of general anesthesia and axillary block on arterial occlusion pressure (AOP) estimation based TP settings in upper limb fracture surgery.

After, ethical committee approval 80 adult patients undergoing upper limb fracture surgery who gave their signed informed consent will be included. The age below 18 and above 85 years, American Society of Anesthesiology (ASA) physical status >2, any contraindication to axillary block or GA, adverse reaction history to anesthetic drugs, severe anemia, and refusal to give informed consent will be the exclusion criteria. The patients will be randomized to one of two study groups using a computer-generated randomization list to receive GA (Group 1) and axillary block (Group 2).

Main endpoints are initial and maximal blood pressures, AOP, initial and maximal TPs, and tourniquet time. Additionally, the surgeon will evaluate the quality of bloodless surgical area with respect to the amount of blood using a 4-point scale (1: Excellent= No blood in the surgical field, 2: Good= Some blood in the surgical field but no interference with surgery, 3: Fair= Blood in the surgical field but no significant interference with surgery, 4: Poor= Blood in the surgical field obscures the view) at the beginning, in the middle, and at the end of the surgical procedure. The patients will be observed for signs of tourniquet related complications by a blind investigator. SPSS 20.0 for Windows is used for data analysis. The t test and the χ2 test will be used for continuous and categorical data respectively. A P value below 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing upper limb fracture surgery

Exclusion Criteria:

* The age below 18 and above 85 years,
* American Society of Anesthesiology (ASA) physical status >2
* Any contraindication to axillary block or general anesthesia
* Any contraindication to tourniquet use
* Adverse reaction history to anesthetic drugs
* Severe anemia
* Refusal to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
Initial and maximal systolic blood pressure (mmHg) | Intraoperative
  Initial and maximal systolic blood pressures define the systolic blood pressures measured and recorded by the patient monitor just before tourniquet inflation and during tourniquet application respectively.
Arterial occlusion pressure (mmHg) | Intraoperative
  Arterial occlusion pressure is the minimal tourniquet pressure required to cease arterial blood flow to the limb and calculated with AOP estimation formula according to initial SBP and Tissue Padding Coefficient (KTP) values (AOP= [SBP+10]/KTP) from a list.
Initial and maximal tourniquet pressures (mmHg) | Intraoperative
  Initial and maximal tourniquet pressures define first adjusted and maximal tourniquet pressures during surgery.
Tourniquet time (minute) | Intraoperative
  Tourniquet time defines the time period between the inflation and deflation of the tourniquet cuff at the beginning and end of the surgery respectively.

SECONDARY OUTCOMES:
The quality of bloodless surgical area | Intraoperative
  The quality of bloodless surgical area will be evaluated by the surgeon respect to the amount of blood using a 4-point scale (1: Excellent= No blood in the surgical field, 2: Good= Some blood in the surgical field but no interference with surgery, 3: Fair= Blood in the surgical field but no significant interference with surgery, 4: Poor= Blood in the surgical field obscures the view) at the beginning, in the middle, and at the end of the surgical procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Estebe JP, Davies JM, Richebe P. The pneumatic tourniquet: mechanical, ischaemia-reperfusion and systemic effects. Eur J Anaesthesiol. 2011 Jun;28(6):404-11. doi: 10.1097/EJA.0b013e328346d5a9. PMID 21502865
- [Background] Odinsson A, Finsen V. Tourniquet use and its complications in Norway. J Bone Joint Surg Br. 2006 Aug;88(8):1090-2. doi: 10.1302/0301-620X.88B8.17668. PMID 16877612
- [Background] Olivecrona C, Blomfeldt R, Ponzer S, Stanford BR, Nilsson BY. Tourniquet cuff pressure and nerve injury in knee arthroplasty in a bloodless field: a neurophysiological study. Acta Orthop. 2013 Apr;84(2):159-64. doi: 10.3109/17453674.2013.782525. Epub 2013 Mar 14. PMID 23485070
- [Background] Olivecrona C, Ponzer S, Hamberg P, Blomfeldt R. Lower tourniquet cuff pressure reduces postoperative wound complications after total knee arthroplasty: a randomized controlled study of 164 patients. J Bone Joint Surg Am. 2012 Dec 19;94(24):2216-21. doi: 10.2106/JBJS.K.01492. PMID 23318611
- [Background] Boya H, Tuncali B, Ozcan O, Arac S, Tuncay C. Practice of tourniquet use in Turkey: a pilot study. Acta Orthop Traumatol Turc. 2016;50(2):162-70. doi: 10.3944/AOTT.2015.15.0066. PMID 26969951
- [Background] Ding L, Ding CY, Wang YL, Wang ML, Qian XH, Huang L, Xie XE, Ji HZ. Application effect of pneumatic tourniquet with individualized pressure setting in orthopaedic surgery of extremities: A meta-analysis. J Adv Nurs. 2019 Dec;75(12):3424-3433. doi: 10.1111/jan.14196. Epub 2019 Oct 15. PMID 31524296
- [Background] Van Roekel HE, Thurston AJ. Tourniquet pressure: the effect of limb circumference and systolic blood pressure. J Hand Surg Br. 1985 Jun;10(2):142-4. doi: 10.1016/0266-7681(85)90002-6. PMID 4031590
- [Background] Pauers RS, Carocci MA. Low pressure pneumatic tourniquets: effectiveness at minimum recommended inflation pressures. J Foot Ankle Surg. 1994 Nov-Dec;33(6):605-9. PMID 7894409
- [Background] Shaw JA, Murray DG. The relationship between tourniquet pressure and underlying soft-tissue pressure in the thigh. J Bone Joint Surg Am. 1982 Oct;64(8):1148-52. PMID 7130227
- [Background] McLaren AC, Rorabeck CH. The pressure distribution under tourniquets. J Bone Joint Surg Am. 1985 Mar;67(3):433-8. PMID 3972869
- [Background] Hargens AR, McClure AG, Skyhar MJ, Lieber RL, Gershuni DH, Akeson WH. Local compression patterns beneath pneumatic tourniquets applied to arms and thighs of human cadavera. J Orthop Res. 1987;5(2):247-52. doi: 10.1002/jor.1100050211. PMID 3572594
- [Background] Graham B, Breault MJ, McEwen JA, McGraw RW. Perineural pressures under the pneumatic tourniquet in the upper extremity. J Hand Surg Br. 1992 Jun;17(3):262-6. doi: 10.1016/0266-7681(92)90111-e. PMID 1624856
- [Background] Estersohn HS, Sourifman HA. The minimum effective midthigh tourniquet pressure. J Foot Surg. 1982 Winter;21(4):281-4. PMID 7186917
- [Background] Newman RJ, Muirhead A. A safe and effective low pressure tourniquet. A prospective evaluation. J Bone Joint Surg Br. 1986 Aug;68(4):625-8. doi: 10.1302/0301-620X.68B4.3525572.
- [Background] Tuncali B, Karci A, Bacakoglu AK, Tuncali BE, Ekin A. Controlled hypotension and minimal inflation pressure: a new approach for pneumatic tourniquet application in upper limb surgery. Anesth Analg. 2003 Nov;97(5):1529-1532. doi: 10.1213/01.ANE.0000081660.97731.91. PMID 14570681
- [Background] Unver B, Karatosun V, Tuncali B. Effects of tourniquet pressure on rehabilitation outcomes in patients undergoing total knee arthroplasty. Orthop Nurs. 2013 Jul-Aug;32(4):217-22. doi: 10.1097/NOR.0b013e31829aef2a. PMID 23881019
- [Background] Tuncali B, Karci A, Tuncali BE, Mavioglu O, Ozkan M, Bacakoglu AK, Baydur H, Ekin A, Elar Z. A new method for estimating arterial occlusion pressure in optimizing pneumatic tourniquet inflation pressure. Anesth Analg. 2006 Jun;102(6):1752-7. doi: 10.1213/01.ane.0000209018.00998.24. PMID 16717321
- [Background] Tuncali B, Boya H, Kayhan Z, Arac S, Camurdan MA. Clinical utilization of arterial occlusion pressure estimation method in lower limb surgery: effectiveness of tourniquet pressures. Acta Orthop Traumatol Turc. 2016;50(2):171-7. doi: 10.3944/AOTT.2015.15.0175. PMID 26969952
- [Background] Tuncali B, Boya H, Kayhan Z, Arac S. Obese patients require higher, but not high pneumatic tourniquet inflation pressures using a novel technique during total knee arthroplasty. Eklem Hastalik Cerrahisi. 2018 Apr;29(1):40-5. doi: 10.5606/ehc.2018.57973. PMID 29526158
- [Background] Tuncali B, Boya H, Kayhan Z, Arac S. Tourniquet pressure settings based on limb occlusion pressure determination or arterial occlusion pressure estimation in total knee arthroplasty? A prospective, randomized, double blind trial. Acta Orthop Traumatol Turc. 2018 Jul;52(4):256-260. doi: 10.1016/j.aott.2018.04.001. Epub 2018 May 8. PMID 29752149
- [Background] Besir A, Tugcugil E. Does Tourniquet Time or Pressure Contribute to Intracranial Pressure Increase following Tourniquet Application? Med Princ Pract. 2019;28(1):16-22. doi: 10.1159/000495110. Epub 2018 Nov 5. PMID 30396181
- [Background] Neal JM, Gerancher JC, Hebl JR, Ilfeld BM, McCartney CJ, Franco CD, Hogan QH. Upper extremity regional anesthesia: essentials of our current understanding, 2008. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):134-70. doi: 10.1097/AAP.0b013e31819624eb. PMID 19282714
- [Background] Bruce BG, Green A, Blaine TA, Wesner LV. Brachial plexus blocks for upper extremity orthopaedic surgery. J Am Acad Orthop Surg. 2012 Jan;20(1):38-47. doi: 10.5435/JAAOS-20-01-038. PMID 22207517
- [Background] Chan VW, Peng PW, Kaszas Z, Middleton WJ, Muni R, Anastakis DG, Graham BA. A comparative study of general anesthesia, intravenous regional anesthesia, and axillary block for outpatient hand surgery: clinical outcome and cost analysis. Anesth Analg. 2001 Nov;93(5):1181-4. doi: 10.1097/00000539-200111000-00025. PMID 11682392
- [Background] Gonano C, Kettner SC, Ernstbrunner M, Schebesta K, Chiari A, Marhofer P. Comparison of economical aspects of interscalene brachial plexus blockade and general anaesthesia for arthroscopic shoulder surgery. Br J Anaesth. 2009 Sep;103(3):428-33. doi: 10.1093/bja/aep173. Epub 2009 Jul 8. PMID 19586958
- [Background] Liu J, Yuan W, Wang X, Royse CF, Gong M, Zhao Y, Zhang H. Peripheral nerve blocks versus general anesthesia for total knee replacement in elderly patients on the postoperative quality of recovery. Clin Interv Aging. 2014 Feb 18;9:341-50. doi: 10.2147/CIA.S56116. eCollection 2014. PMID 24600214
- [Background] Bergmann I, Heetfeld M, Crozier TA, Schafdecker HG, Pöschl R, Wiese CH, et al. Peripheral nerve blocks give greater hemodynamic stability than general anesthesia for ASA III patients undergoing outpatient knee arthroscopy. Cent Eur J Med 2013; 8:436-42.
- [Background] Harsanji Drenjancevic I, Drenjancevic D, Davidovic-Cvetko E, Drenjancevic I, Gulam D, Kvolik S. DOES THE ANESTHESIA TECHNIQUE AFFECT ARTERIAL PRESSURE AND REGIONAL CEREBRAL OXYGEN SATURATION DURING SHOULDER ARTHROSCOPY IN THE BEACH CHAIR POSITION? Acta Clin Croat. 2018 Sep;57(3):473-479. doi: 10.20471/acc.2018.57.03.10. PMID 31168180
- [Background] Ozzeybek D, Oztekin S, Mavioglu O, Karaege G, Ozkardesler S, Ozkan M, Canyilmaz M, Elar Z. Comparison of the haemodynamic effects of interscalene block combined with general anaesthesia and interscalene block alone for shoulder surgery. J Int Med Res. 2003 Sep-Oct;31(5):428-33. doi: 10.1177/147323000303100512. PMID 14587312
- [Background] Crenshaw AG, Hargens AR, Gershuni DH, Rydevik B. Wide tourniquet cuffs more effective at lower inflation pressures. Acta Orthop Scand. 1988 Aug;59(4):447-51. doi: 10.3109/17453678809149401. PMID 3421083
- [Background] Younger AS, McEwen JA, Inkpen K. Wide contoured thigh cuffs and automated limb occlusion measurement allow lower tourniquet pressures. Clin Orthop Relat Res. 2004 Nov;(428):286-93. doi: 10.1097/01.blo.0000142625.82654.b3. PMID 15534554
- [Background] Mittal P, Shenoy S, Sandhu JS. Effect of different cuff widths on the motor nerve conduction of the median nerve: an experimental study. J Orthop Surg Res. 2008 Jan 9;3:1. doi: 10.1186/1749-799X-3-1. PMID 18182119
- [Background] Kovar FM, Jaindl M, Oberleitner G, Endler G, Breitenseher J, Prayer D, Kasprian G, Kutscha-Lissberg F. Nerve compression and pain in human volunteers with narrow vs wide tourniquets. World J Orthop. 2015 May 18;6(4):394-9. doi: 10.5312/wjo.v6.i4.394. eCollection 2015 May 18. PMID 25992317